CLINICAL TRIAL: NCT02038829
Title: A Dose-Range Finding Study of SUN-101 in Subjects With Moderate to Severe COPD: GOLDEN 6 (Glycopyrrolate for Obstructive Lung Disease Via Electronic Nebulizer)
Brief Title: A Dose-Range Finding Study of SUN-101 in Subjects With Moderate to Severe COPD
Acronym: GOLDEN 6
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sunovion Respiratory Development Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SUN101-201
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Results first posted 2018-01-25 (Actual); Last update posted 2018-04-10 (Actual); Status verified 2018-03

CONDITIONS: COPD
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): Placebo bid
  Interventions: Drug: Placebo
- SUN-101 3 mcg (Experimental): SUN-101 3 mcg bid
  Interventions: Drug: SUN101 3 mcg
- SUN-101 6.25 mcg (Experimental): SUN-101 6.25 mcg bid
  Interventions: Drug: SUN-101 6.25 mcg
- SUN-101 12.5 mcg (Experimental): SUN-101 12.5 mcg bid
  Interventions: Drug: SUN-101 12.5 mcg
- SUN-101 50 mcg (Experimental): SUN-101 50 mcg bid
  Interventions: Drug: SUN-101 50 mcg
- Aclidinium 400 mcg (Active Comparator): Aclidinium 400 mcg bid
  Interventions: Drug: Aclidinium

INTERVENTIONS:
Drug: Placebo — Placebo
  Arms: Placebo
Drug: SUN101 3 mcg — SUN-101 3 mcg bid
  Arms: SUN-101 3 mcg
Drug: SUN-101 6.25 mcg — SUN-101 6.25 mcg bid
  Arms: SUN-101 6.25 mcg
Drug: SUN-101 12.5 mcg — SUN-101 12.5 mcg bid
  Arms: SUN-101 12.5 mcg
Drug: SUN-101 50 mcg — SUN-101 50 mcg bid
  Arms: SUN-101 50 mcg
Drug: Aclidinium — Aclidinium 400 mcg bid
  Arms: Aclidinium 400 mcg

SUMMARY:
Study for subjects 40 to 65 years-old with a diagnosis of moderate to severe COPD. Aclidinium bromide 400 mcg 2x a day will be given as an active comparator.

DETAILED DESCRIPTION:
This is a randomized, six-way crossover study to determine the efficacy and dose-response profile of SUN101. The study population will consist of subjects 40 to 65 years-old (inclusive), with a diagnosis of moderate to severe COPD. Aclidinium bromide 400 mcg bid will be given as an active comparator. The study will be double-blind for SUN-101 and placebo and will be open-label for aclidinium.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 40 to 65 years-old, inclusive.
2. A clinical diagnosis of moderate to severe COPD according to the GOLD 2011 guidelines.
3. Current smokers or ex-smokers with at least 10 pack year smoking history (eg, at least 1 pack/day for 10 years, or equivalent).
4. Post bronchodilator (following inhalation of ipratropium bromide) FEV1 ≥ 40% and ≤ 70% of predicted normal during Screening.
5. Post bronchodilator (following inhalation of ipratropium bromide) FEV1/FVC ratio ≤ 0.70 during Screening.
6. Post bronchodilator (following inhalation of ipratropium bromide) improvement in FEV1 ≥ 12% and ≥ 100 mL during Screening.
7. Ability to perform reproducible spirometry according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines (2005).
8. Female of child bearing potential (only) must have a negative serum pregnancy test at Screening and be neither breastfeeding nor intending to become pregnant during study participation. Females of childbearing potential must be instructed to and agree to avoid pregnancy during the study. Female subjects of child bearing potential must use an adequate method of birth control from Screening until 30 days after receiving study drug and use contraception in addition to their partners using a barrier method. Acceptable forms of contraception are as follows:

   * Abstinence
   * Barrier methods: condoms, diaphragms, cervical caps; with a spermicide foam, gel, film, cream or suppository;
   * Oral contraceptives
   * Non hormone containing intrauterine methods: intrauterine devices or systems.
9. Willing and able to remain at the study site for at least 24 hours at Day 7 of each Treatment Period.
10. Willing and able to attend all study visits and adhere to all study assessments/procedures.
11. Willing and able to provide written informed consent

Exclusion Criteria:

1. Current evidence or recent history of any clinically significant and unstable disease (other than COPD) or abnormality in the opinion of the Investigator that would put the subject at risk or which would compromise the quality of the study data; including but not limited to cardiovascular disease, myocardial infarction, cardiac failure, uncontrolled hypertension, life threatening arrhythmias, uncontrolled diabetes, neurologic or neuromuscular disease, liver disease, gastrointestinal disease or electrolyte abnormalities.
2. Current evidence or history of a clinically significant abnormality of cardiac rhythm and/or conduction including Holter monitoring prior to randomization.
3. Primary diagnosis of asthma.
4. History of malignancy of any organ system, treated or untreated within the past 5 years, with the exception of localized basal cell carcinoma of the skin.
5. Recent history of COPD exacerbation requiring hospitalization or need for increased treatments for COPD within 6 weeks prior to Screening.
6. Use of daily oxygen therapy > 10 hours per day.
7. Use of systemic steroids within 3 months prior to Screening.
8. Respiratory tract infection within 6 weeks prior to or during Screening.
9. History of tuberculosis, bronchiectasis or other non-specific pulmonary disease.
10. History of urinary retention or bladder neck obstruction type symptoms.
11. History of narrow angle glaucoma.
12. Prolonged QTcF interval (males > 450 msec and females >470 msec) during Screening, or history of long QT syndrome.
13. Recent history (previous 12 months) of excessive use or abuse of alcohol or narcotic/illegal drugs.
14. History of hypersensitivity or intolerance to aerosol medications, beta-2 agonists, or anticholinergics.
15. Participation in another investigational drug study where drug was received within 30 days prior to Screening, or current participation in another investigational drug trial.
16. Subject is a staff member of the clinical site or a relative of a clinical site staff member.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2014-01; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: SUN101 Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (10):
- United States (10):
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - American Health Research, Inc., Charlotte, North Carolina
  - North Carolina Clinical Research, Raleigh, North Carolina
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Palmetto Medical Research Associates, LLC, Easley, South Carolina
  - Greenville Pharmaceutical Research, Inc., Greenville, South Carolina
  - Upstate Pharmaceutical Research, Greenville, South Carolina
  - S. Carolina, Spartanburg, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - CU Pharmaceutical Research, Union, South Carolina

REFERENCES:
- [Result] Donohue JF, Goodin T, Tosiello R, Wheeler A. Dose selection for glycopyrrolate/eFlow(R) phase III clinical studies: results from GOLDEN (Glycopyrrolate for Obstructive Lung Disease via Electronic Nebulizer) phase II dose-finding studies. Respir Res. 2017 Dec 4;18(1):202. doi: 10.1186/s12931-017-0681-z. PMID 29202767

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Eligible subjects will be randomized to one of 12 treatment sequences. There will be a minimum of a 7-day washout period between each treatment visit. At each visit, subjects will receive one dose of study medication according to the sequence assigned.
Groups:
- Treatment Group 1: Participants received SUN-101 50mcg; Aclidinium 400mcg; Placebo; SUN-101 6,25mcg; SUN-101 3mcg; SUN-101 12.5mcg
- Treatment Group 2: Participants received Placebo; SUN-101 50mcg; SUN-101 3mcg Aclidinium 400mcg; SUN-101 12.5 mcg; SUN-101 6mcg
- Treatment Group 3: Participants received SUN-101 3mcg Placebo; SUN-101 12.5 mcg; SUN-101 50mcg; SUN-101 6.25mcg Aclidinium 400mcg;
- Treatment Group 4: Participants received SUN-101 12.5 mcg; SUN-101 3mcg Placebo; SUN-101 50mcg; Aclidinium 400mcg; SUN-101 6.25mcg
- Treatment Group 5: Participants received SUN-101 6.25mcg SUN-101 12.5 mcg; Aclidinium 400mcg; SUN-101 3mcg SUN-101 50mcg Placebo;
  Aclidinium 400mcg; SUN-101 6.25mcg
- Treatment Group 6: Participants received Aclidinium 400mcg; SUN-101 6.25mcg SUN-101 50mcg SUN-101 12.5 mcg; Placebo; SUN-101 3mcg
  Placebo;
- Treatment Group 7: Participants received SUN-101 3mcg SUN-101 50mcg Aclidinium 400mcg; Placebo; SUN-101 6.25mcg SUN-101 12.5 mcg;
  SUN-101 3mcg
- Treatment Group 8: Participants received Aclidinium 400mcg; SUN-101 3mcg SUN-101 6.25mcg SUN-101 50mcg SUN-101 12.5 mcg; Placebo;
- Treatment Group 9: Participants received SUN-101 6.25mcg Aclidinium 400mcg; SUN-101 12.5 mcg SUN-101 3mcg Placebo; SUN-101 50mcg
- Treatment Group 10: Participants received SUN-101 12.5 mcg SUN-101 6.25mcg Placebo; Aclidinium 400mcg; SUN-101 50 mcg SUN-101 3mcg
- Treatment Group 11: Participants received Placebo; SUN-101 12.5 mcg SUN-101 50 mcg SUN-101 6.25mcg Aclidinium 400mcg; SUN-101 3mcg
- Treatment Group 12: Participants received SUN-101 50 mcg Placebo; SUN-101 3mcg SUN-101 6.25mcg Aclidinium 400mcg; SUN-101 12.5 mcg
Period: Treatment Period 1
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 1
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 2
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 8 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 8 | 8
Completed | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 8
Not Completed | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 2
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 8 | 8 | 8 | 7 | 8 | 8 | 8 | 8 | 8 | 7 | 8
Completed | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 3
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 3
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 4
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 8 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 7 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 4
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 7 | 8 | 8 | 7 | 7 | 8 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 5
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout Period 5
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Treatment Period 6
Arm/Group | Treatment Group 1 | Treatment Group 2 | Treatment Group 3 | Treatment Group 4 | Treatment Group 5 | Treatment Group 6 | Treatment Group 7 | Treatment Group 8 | Treatment Group 9 | Treatment Group 10 | Treatment Group 11 | Treatment Group 12
Started | 7 | 7 | 8 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Completed | 7 | 7 | 7 | 8 | 7 | 7 | 7 | 8 | 7 | 8 | 7 | 8
Not Completed | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all participants
Arm/Group | Total
Number analyzed (Participants) | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 94
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (5.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 46
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 96
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 86
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 96

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Trough FEV1 at Treatment Visit Day 7 Compared to Placebo.
Description: Spirometry was performed according to internationally accepted standards. Trough FEV1 was defined as the average of the 2 spirometry values collected at 23 hours 15 minutes, and 23 hours 45 minutes post-morning dose on Day 7 of each Treatment Period. The FEV1 values within 6 hours after the use of rescue medication were considered as missing. Baseline was calculated as the mean of the FEV1 values at 45 minutes and 15 minutes prior to the morning dose at Day 1 of each Treatment Period
Time Frame: Baseline and Day 7
Population: Efficacy Population: all subjects who were randomized to treatment, received at least one dose of study medication, and had at least one trough FEV1 evaluation and the corresponding baseline FEV1 for at least one treatment period.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo | SUN-101 3 mcg | SUN-101 6.25 mcg | SUN-101 12.5 mcg | SUN-101 50 mcg | Aclidinium 400 mcg
Number analyzed (Participants) | 92 | 91 | 92 | 90 | 92 | 94
liters | -0.0282 (0.0300) | -0.0156 (0.0300) | 0.0540 (0.0238) | 0.0806 (0.0300) | 0.1092 (0.0300) | 0.1285 (0.0300)
Statistical Analysis 1: Comparison: Placebo vs SUN-101 3 mcg; An mixed effects model was used with mean change from baseline in trough FEV1 as the response, with factors for treatment, period, sequence, baseline FEV1 as a covariate and a random effect for subject nested within sequence. The Kenward and Roger correction to the degrees of freedom was used. An unstructured covariance model was used to model intrasubject correlation; Test type: Superiority — A sample size of 66 subjects (rounding to 72 for using Williams squares and 96 with dropouts) provides ~90% power to detect a 100 mL treatment difference in mean change trough FEV1 between SUN-101 and placebo at a Bonferroni-adjusted significance level of 0.0125 using a 2-tailed paired t-test and assuming a within-subject standard deviation for change in trough FEV1 of 176 and a within-subject correlation of 0.3; p = 0.9730, LS Mean (SE) — P-values were adjusted using Dunnett's method for comparing the multiple treatments to placebo. The comparison of aclidinium to placebo was performed at the 0.05 significance level to establish assay sensitivity; LS Mean (SE) = 0.0126, 95% CI 2-sided [-0.0318 to 0.0569], Standard Error of Mean 0.0225
Statistical Analysis 2: Comparison: Placebo vs SUN-101 6.25 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p = 0.0014, LS Mean (SE) — [p-value comment as in outcome 1, analysis 1]; LS Mean (SE) = 0.0822, 95% CI 2-sided [0.0380 to 0.1264], Standard Error of Mean 0.0225
Statistical Analysis 3: Comparison: Placebo vs SUN-101 12.5 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, LS Mean (SE) — [p-value comment as in outcome 1, analysis 1]; LS Mean (SE) = 0.1088, 95% CI 2-sided [0.0644 to 0.1532], Standard Error of Mean 0.0226
Statistical Analysis 4: Comparison: Placebo vs SUN-101 50 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, LS Mean (SE) — [p-value comment as in outcome 1, analysis 1]; LS Mean (SE) = 0.1375, 95% CI 2-sided [0.0931 to 0.1818], Standard Error of Mean 0.0226
Statistical Analysis 5: Comparison: Placebo vs Aclidinium 400 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority — [test comment as in outcome 1, analysis 1]; p < 0.0001, LS Mean (SE) — [p-value comment as in outcome 1, analysis 1]; LS Mean (SE) = 0.1567, 95% CI 2-sided [0.1121 to 0.2012], Standard Error of Mean 0.0226

2. Secondary Outcome: Standardized Change From Baseline in FEV1 AUC(0-12hours)
Description: The standardized FEV1 AUC(0-12) on Day 7 was calculated using the trapezoidal rule from the changes in FEV1 from the baseline value (the mean of the two FEV1 values at 45 minutes and 15 minutes prior to morning dose at Day 1 of the respective Treatment Periods) and dividing by the actual length of the time interval).
Time Frame: Day 7
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | Placebo | SUN-101 3 mcg | SUN-101 6.25 mcg | SUN-101 12.5 mcg | SUN-101 50 mcg | Aclidinium 400 mcg
Number analyzed (Participants) | 92 | 91 | 92 | 90 | 92 | 94
Liters | -0.0203 (0.0315) | 0.0323 (0.0316) | 0.0639 (0.0315) | 0.1052 (0.0316) | 0.1760 (0.0315) | 0.1699 (0.0316)
Statistical Analysis 1: Comparison: Placebo vs SUN-101 3 mcg; An mixed effects model was used with standardized FEV1 AUC(0-12) on Day 7 as the response, with factors for treatment, period, sequence, baseline FEV1 as a covariate and a random effect for subject nested within sequence. The Kenward and Roger correction to the degrees of freedom was used. An unstructured covariance model was used to model intrasubject correlation; Test type: Superiority — A sample size of 78 subjects (rounding to 84 for using Williams squares) provides ~80% power to detect a 55 mL treatment difference in mean change trough FEV1 between SUN-101 and placebo at a Bonferroni-adjusted significance level of 0.0125 using a 2-tailed paired t-test and assuming a within-subject standard deviation for change in AUC(0-12) of 143 and a within-subject correlation of 0.3; p = 0.0046, LS Mean (SE); LS Mean (SE) = 0.0526, 95% CI 2-sided [0.0163 to 0.0888], Standard Error of Mean 0.0184
Statistical Analysis 2: Comparison: Placebo vs SUN-101 6.25 mcg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, LS Mean (SE); LS Mean (SE) = 0.0842, 95% CI 2-sided [0.0478 to 0.1206], Standard Error of Mean 0.0185
Statistical Analysis 3: Comparison: Placebo vs SUN-101 12.5 mcg; [analysis description as in outcome 2, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, LS Mean (SE); LS Mean (SE) = 0.1255, 95% CI 2-sided [0.0890 to 0.1621], Standard Error of Mean 0.0186
Statistical Analysis 4: Comparison: Placebo vs SUN-101 50 mcg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, LS Mean (SE); LS Mean (SE) = 0.1963, 95% CI 2-sided [0.1601 to 0.2325], Standard Error of Mean 0.0184
Statistical Analysis 5: Comparison: Placebo vs Aclidinium 400 mcg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — [test comment as in outcome 2, analysis 1]; p < 0.0001, LS Mean (SE); LS Mean (SE) = 0.1902, 95% CI 2-sided [0.1537 to 0.2268], Standard Error of Mean 0.0186

3. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (Overall and by Treatment)
Description: A treatment emergent adverse event (TEAE) is any TEAE that occurred on or after the first dose of study medication, any SAE with a missing start date and a stop date on or after the first dose of study medication, or any TEAE with both a missing start and stop date.
Time Frame: Over 7 days
Population: Safety population was defined as all subjects who were randomized to treatment and received at least one dose of study medication.
Measure: Number; unit: participants
Groups:
- TOTAL: Total number of study participants
Arm/Group | Placebo | SUN-101 3 mcg | SUN-101 6.25 mcg | SUN-101 12.5 mcg | SUN-101 50 mcg | Aclidinium 400 mcg | TOTAL
Number analyzed (Participants) | 92 | 91 | 92 | 90 | 92 | 94 | 96
participants | 11 | 22 | 23 | 24 | 14 | 24 | 62

4. Secondary Outcome: Percentage of Subjects With Treatment-emergent Adverse Events (Overall and by Treatment)
Description: as for outcome 3
Time Frame: Over 7 days
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | SUN-101 3 mcg | SUN-101 6.25 mcg | SUN-101 12.5 mcg | SUN-101 50 mcg | Aclidinium 400 mcg | TOTAL
Number analyzed (Participants) | 92 | 91 | 92 | 90 | 92 | 94 | 96
percentage of participants | 12.0 | 24.2 | 25.0 | 26.7 | 15.2 | 25.5 | 64.6

ADVERSE EVENTS:
Time Frame: Over 7 days
Description: A treatment emergent serious adverse event (TESAE) is any SAE that occurred on or after the first dose of study medication, any SAE with a missing start date and a stop date on or after the first dose of study medication, or any SAE with both a missing start and stop date.
Arm/Group | Placebo | SUN-101 3 mcg | SUN-101 6.25 mcg | SUN-101 12.5 mcg | SUN-101 50 mcg | Aclidinium 400 mcg
Serious Adverse Events (participants affected / at risk) | 1/92 | 0/91 | 2/92 | 1/90 | 0/92 | 3/94
Other Adverse Events (participants affected / at risk) | 2/92 | 6/91 | 4/92 | 6/90 | 5/92 | 10/94
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | SUN-101 3 mcg (N=91) | SUN-101 6.25 mcg (N=92) | SUN-101 12.5 mcg (N=90) | SUN-101 50 mcg (N=92) | Aclidinium 400 mcg (N=94)
acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
cardia failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
metapneumovirus infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 | 1 (1)
pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=92) | SUN-101 3 mcg (N=91) | SUN-101 6.25 mcg (N=92) | SUN-101 12.5 mcg (N=90) | SUN-101 50 mcg (N=92) | Aclidinium 400 mcg (N=94)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 8 (8)
cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 6 (6) | 3 (3) | 6 (6) | 4 (4) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.